CLINICAL TRIAL: NCT00607724
Title: An Open-Label, Phase I Study of Systemic Hedgehog Pathway Antagonist, GDC-0449, in Patients With Locally Advanced or Metastatic Solid Tumors That Are Refractory to Standard Therapy or For Whom No Standard Therapy Exists
Brief Title: GDC-0449 in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000585468; JHOC-J06131; GENETECH-SHH3925g; NCT00862771 (obsolete NCT alias)
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — HhAntag691

ARMS (7):
- Stage 1: GDC-0449 (150 mg) (Experimental): Participants with any tumor received a single oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 milligram (mg) on Day 1. Beginning on Day 8, participants received once daily doses of GDC-0449 150 mg, orally, continuing until disease progression (deterioration of evaluable lesions and/or tumor-related symptoms defined using Response Evaluation Criteria in Solid Tumors Version 1.0 (RECIST v1.0), maximum benefit, or intolerability.
  Interventions: Drug: GDC-0449
- Stage 1: GDC-0449 (270 mg) (Experimental): Participants with any tumor received a single oral dose of GDC-0449 hard gelatin capsules at a dosage of 270 mg on Day 1. Beginning on Day 8, participants received once daily doses of GDC-0449 270 mg, orally, continuing until disease progression, maximum benefit, or intolerability.
  Interventions: Drug: GDC-0449
- Stage 1: GDC-0449 (540 mg) (Experimental): Participants with any tumor received a single oral dose of GDC-0449 hard gelatin capsules at a dosage of 540 mg on Day 1. Beginning on Day 8, participants received once daily doses of GDC-0449 540 mg, orally, continuing until disease progression, maximum benefit, or intolerability.
  Interventions: Drug: GDC-0449
- Stage 2: BCC [GDC-0449 (150 mg)] (Experimental): Participants with basal cell carcinoma (BCC) received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
  Interventions: Drug: GDC-0449
- Stage 2: BCC [GDC-0449 (270 mg)] (Experimental): Participants with BCC received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 270 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
  Interventions: Drug: GDC-0449
- Stage 2:Safety Expansion Cohort [GDC-0449 (150 mg)] (Experimental): Participants received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
  Interventions: Drug: GDC-0449
- Stage 2: New Formulation [GDC-0449 (150 mg )] (Experimental): Participants received a daily oral dose of GDC-0449 Phase II drug product hard gelatin capsules at a dosage of 150 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
  Interventions: Drug: GDC-0449

INTERVENTIONS:
Drug: GDC-0449
  Other Names: Hedgehog Pathway Inhibitor

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as GDC-0449, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of GDC-0449 in treating patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and tolerability of escalating doses of systemic Hedgehog antagonist GDC-0449 in patients with locally advanced or metastatic solid tumors.
* To estimate the maximum tolerated dose of GDC-0449 in these patients.
* To define the dose-limiting toxicities of GDC-0449 in these patients.
* To characterize the pharmacokinetic properties of GDC-0449 following a single dose and multiple doses.
* To determine the recommended phase II dose and schedule of GDC-0449 for efficacy testing based on achievement of the target exposure with an acceptable safety profile.

Secondary

* To determine whether inhibition of Hedgehog (Hh) signaling by GDC-0449 can be reliably measured in human hair follicles and to define the relationship between this pharmacodynamic (PD) effect in surrogate tissue and GDC-0449 dose and exposure.
* To make a preliminary assessment of tumor response in patients treated with this drug.

Tertiary

* To examine modulation of Hh target genes (other than GLI1) by GDC-0449 in hair follicles and/or tumor tissue.

OUTLINE: This is a multicenter study.

Patients receive oral systemic Hedgehog antagonist GDC-0449 once on day 1 and then once or twice daily beginning on day 8 and continuing for up to 49 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo plasma, urine, and hair sample collection and skin punch biopsies periodically for pharmacokinetic and pharmacodynamic analyses. The plasma and urine samples are analyzed separately using liquid chromatography/tandem mass spectrometry-based methods. Ex vivo plasma protein binding of GDC-0449 is assayed using an equilibrium dialysis approach. Expression levels of Gli1 and other Hedgehog target genes in hair follicle samples and/or tumor tissue are measured at the RNA level using qRT-PCR.

After completion of study therapy, patients are followed at 21 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally advanced or metastatic solid tumor that is refractory to standard therapy or for which no standard therapy exists

  * Progressed after first-line and second-line therapy (if there is a second-line therapy that has been shown to provide clinical benefit)

    * Must receive standard second-line therapy if second-line therapy has been shown to provide clinical benefit
* Evaluable disease by physical examination, imaging, and/or one of the following:

  * Two rising prostate-specific antigen (PSA) levels ≥ 2 weeks apart, with one obtained during screening (for patients with prostate cancer)
  * Two rising CA-125 levels ≥ 2 weeks apart, with one obtained during screening (for patients with ovarian cancer)
* No CNS cancer, either primary lesions or metastatic disease, as the current malignancy
* No pleural effusions, ascites, or leptomeningeal disease as the only manifestation of the current malignancy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Granulocyte count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Serum bilirubin normal
* Alkaline phosphatase ≤ 1.5 times upper limit of normal (ULN) (≤ 4 times ULN for patients with liver or bone metastases)
* AST and ALT ≤ 1.5 times ULN (≤ 5 times the ULN for patients with liver metastases)
* Serum creatinine ≤ 1.5 mg/dL
* INR < 1.3
* aPTT ≤ 1.5 times ULN
* Fasting total serum cholesterol ≤ 220 mg/dL (without cholesterol-lowering drugs)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able and willing to swallow pills
* No malabsorption syndrome or other condition that would interfere with enteral absorption
* No history of significant atherosclerotic disease, including the following:

  * Coronary artery disease (i.e., myocardial infarction within the past year or unstable angina)
  * Documented carotid atheromas
* No history of congestive heart failure or ventricular arrhythmia requiring medication
* No congenital long QT syndrome
* No baseline QTc intervals > 0.47 seconds on two of three baseline 12-lead ECGs recorded during the screening period
* No active infection requiring intravenous antibiotics
* No known HIV infection
* No uncontrolled hypocalcemia, hypomagnesemia, or hypokalemia, defined as less than the lower limit of normal for the institution despite adequate electrolyte supplementation
* No history of clinically important liver disease, including cirrhosis or viral or other hepatitis
* No current alcohol abuse
* No significant traumatic injury within the past 3 weeks
* No other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the study results or renders the patient at high risk from treatment complications

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy, investigational therapy, radiotherapy, or major surgical procedure and recovered
* No concurrent medications with narrow therapeutic indices that are cytochrome P450 substrates (warfarin sodium [Coumadin®])
* No concurrent medications known to prolong the QT interval, including any of the following:

  * Quinidine or other anti-arrhythmic agents
  * Haloperidol, fluoxetine, paroxetine, or sertraline
  * Pentamidine, fluoroquinolone, or macrolide antibiotics
* No concurrent medications that may interfere with the metabolism of GDC-0449 (e.g., ketoconazole)
* No concurrent grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

REFERENCES:
- [Derived] Thacker CA, Weiss GJ, Tibes R, Blaydorn L, Downhour M, White E, Baldwin J, Hoff DD, Korn RL. 18-FDG PET/CT assessment of basal cell carcinoma with vismodegib. Cancer Med. 2012 Oct;1(2):230-6. doi: 10.1002/cam4.33. Epub 2012 Sep 17. PMID 23342272
- [Derived] Von Hoff DD, LoRusso PM, Rudin CM, Reddy JC, Yauch RL, Tibes R, Weiss GJ, Borad MJ, Hann CL, Brahmer JR, Mackey HM, Lum BL, Darbonne WC, Marsters JC Jr, de Sauvage FJ, Low JA. Inhibition of the hedgehog pathway in advanced basal-cell carcinoma. N Engl J Med. 2009 Sep 17;361(12):1164-72. doi: 10.1056/NEJMoa0905360. Epub 2009 Sep 2. PMID 19726763

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)]: Participants with basal cell carcinoma (BCC) received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
- Stage 2: Basal Cell Carcinoma [GDC-0449 (270 mg)]: Participants with BCC received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 270 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
Period: Stage 1: Dose Escalation
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)] | Stage 2: Basal Cell Carcinoma [GDC-0449 (270 mg)] | Stage 2:Safety Expansion Cohort [GDC-0449 (150 mg)] | Stage 2: New Formulation [GDC-0449 (150 mg )]
Started | 7 | 9 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 1 (Participants still on treatment at time of study closure were considered 'completers'.) | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 8 | 4 | 0 | 0 | 0 | 0
Not completed — Tumour Progression-Clinical/Radiographic | 7 | 8 | 4 | 0 | 0 | 0 | 0
Period: Stage 2: Expanded Cohort
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)] | Stage 2: Basal Cell Carcinoma [GDC-0449 (270 mg)] | Stage 2:Safety Expansion Cohort [GDC-0449 (150 mg)] | Stage 2: New Formulation [GDC-0449 (150 mg )]
Started | 0 | 0 | 0 | 6 | 14 | 12 | 16
Completed | 0 | 0 | 0 | 1 (Participants still on treatment at time of study closure were considered 'completers'.) | 5 (Participants still on treatment at time of study closure were considered 'completers'.) | 0 | 5 (Participants still on treatment at time of study closure were considered 'completers'.)
Not Completed | 0 | 0 | 0 | 5 | 9 | 12 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Tumour Progression-Clinical/Radiographic | 0 | 0 | 0 | 4 | 8 | 11 | 10
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety-evaluable population included all participants who received any amount of GDC-0449.
Groups:
- Stage 1: GDC-0449 (150 mg): Participants with any tumor received a single oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 mg on Day 1. Beginning on Day 8, participants received once daily doses of GDC-0449 150 mg, orally, continuing until disease progression, maximum benefit, or intolerability.
- Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)]: Participants with BCC received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
- Total: Total of all reporting groups
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)] | Stage 2: Basal Cell Carcinoma [GDC-0449 (270 mg)] | Stage 2:Safety Expansion Cohort [GDC-0449 (150 mg)] | Stage 2: New Formulation [GDC-0449 (150 mg )] | Total
Number analyzed (Participants) | 7 | 9 | 4 | 6 | 14 | 12 | 16 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.5) | 59.9 (12.6) | 42.3 (15.3) | 54.2 (15.3) | 54.7 (11.2) | 55.3 (14.8) | 54.6 (11.0) | 55.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 1 | 1 | 4 | 5 | 6 | 24
  Male | 5 | 4 | 3 | 5 | 10 | 7 | 10 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any Grade 3 or 4 hematologic or major organ toxicity as graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 3.0) that occurred during the first 35 days after the initiation of study drug (Days 1-35) and was attributable to GDC-0449.
Time Frame: Up to Week 6
Population: Safety-evaluable population.
Measure: Number; unit: percentage of participants
Groups:
- Stage 2: Basal Cell Carcinoma (GDC-0449 [150 mg]): Participants with BCC received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
- Stage 2: Basal Cell Carcinoma (GDC-0449 [270 mg]): Participants with BCC received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 270 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
- Stage 2:Safety Expansion Cohort (GDC-0449 [150 mg]): Participants received a daily oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
- Stage 2: New Formulation (GDC-0449 [150 mg]): Participants received GDC-0449 Phase II drug product as 150-mg hard gelatin capsules daily, orally, starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma (GDC-0449 [150 mg]) | Stage 2: Basal Cell Carcinoma (GDC-0449 [270 mg]) | Stage 2:Safety Expansion Cohort (GDC-0449 [150 mg]) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 7 | 9 | 4 | 6 | 14 | 12 | 16
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) After a Single Dose of GDC-0449
Description: Phase I comprised of two stages, a dose-escalation stage with the goal of estimating the maximum tolerated dose (Stage 1), and an expanded cohort to collect additional safety, PK, and pharmacodynamic (PD) data at the proposed Phase II dose (Stage 2). Phase II represented the additional cohort initiated with 150 mg hard gelatin capsule identified from the safety, PK and PD data from Stage 1 of the trial.
Time Frame: -5 minutes (pre-dose) and 0.5, 1, 2, 4, 8, 24 hours post-dose on Day 1; additionally for stage 1 arms: 48 hours (Day 3), 72 hours (Day 4) post-dose and - 5 minutes (pre-dose) on Day 8
Population: Pharmacokinetic (PK)-evaluable population included participants who had at least Day 1 PK samples available.
Measure: Mean (Standard Deviation); unit: micromolar (mcM)
Groups:
- Stage 2: New Formulation (GDC-0449 [150 mg]): Participants received a daily oral dose of GDC-0449 Phase II drug product hard gelatin capsules at a dosage of 150 mg starting on Day 1 and continuing until disease progression, maximum benefit, or intolerability.
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 7 | 9 | 4 | 16
micromolar (mcM)
  Phase I | 3.58 (1.34) | 6.34 (3.40) | 6.81 (2.69) | NA (NA) — The arm was only valid for Phase II.
  Phase II | NA (NA) — The arm was only valid for Phase I. | NA (NA) — The arm was only valid for Phase I. | NA (NA) — The arm was only valid for Phase I. | 7.2 (3.38)

3. Primary Outcome: Cmax After Multiple Doses of GDC-0449
Description: Cmax was estimated if there were extensive PK sampling in more that 50% of the participants to form a curve.
Time Frame: -5 minutes (pre-dose), 0.5,1,2,4,8 hours post-dose on Day [D] 1; 2,3,4; -5 minutes (pre-dose) on D8,15,22,29,36,64,92,120,148,176,204,232,260,288,316,344;every 4 weeks after D345; end of treatment and study (up to 28 days after last dose), up to 2 years
Population: Cmax was not reported as there were <50% participants with extensive PK sampling and the PK profiles were flat over 24 hours at steady state which did not allow estimation of Cmax.
Groups:
- Stage 1+Stage 2: GDC-0449 (150 mg): Participants with any tumor or BCC or safety expansion cohort received single or daily oral dose of GDC-0449 hard gelatin capsules at 150 mg starting on Day 1 (Stage 1 and Stage 2) and/or Day 8 (Stage 1), until disease progression, maximum benefit, or intolerability.
- Stage 1+Stage 2: GDC-0449 (270 mg): Participants with any tumor or BCC or safety expansion cohort received single or daily oral dose of GDC-0449 hard gelatin capsules at 270 mg starting on Day 1 (Stage 1 and Stage 2) and/or Day 8 (Stage 1), until disease progression, maximum benefit, or intolerability.
Arm/Group | Stage 1+Stage 2: GDC-0449 (150 mg) | Stage 1+Stage 2: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg)
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) After a Single Dose of GDC-0449
Description: Phase I comprised of two stages, a dose-escalation stage with the goal of estimating the maximum tolerated dose (Stage 1), and an expanded cohort to collect additional safety, PK, and PD data at the proposed Phase II dose (Stage 2). Phase II represented the additional cohort initiated with 150 mg hard gelatin capsule identified from the safety, PK and PD data from Stage 1 of the trial.
Time Frame: as for outcome 2
Population: PK-evaluable population.
Measure: Median (Full Range); unit: days
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 7 | 9 | 4 | 16
days
  Phase I | 2 [0.0417 to 7] | 2 [1 to 3] | 2.5 [0.167 to 3] | NA [NA to NA] — The arm was only valid for Phase II.
  Phase II | NA [NA to NA] — The arm was only valid for Phase I. | NA [NA to NA] — The arm was only valid for Phase I. | NA [NA to NA] — The arm was only valid for Phase I. | 1 [0.0833 to 1]

5. Primary Outcome: Tmax After Multiple Doses of GDC-0449
Description: Tmax was estimated if there were extensive PK sampling in more that 50% of the participants to form a curve.
Time Frame: as for outcome 3
Population: Cmax was not reported as there were <50% participants with extensive PK sampling and the PK profiles were flat over 24 hours at steady state which did not allow estimation of Cmax, and as Tmax was related to Cmax, it was also not estimated.
Groups:
- Stage 1+Stage 2: GDC-0449 (270 mg): Participants with any tumor or BCC or safety expansion cohort received single or daily oral dose of GDC-0449 hard gelatin capsules at 150 mg starting on Day 1 (Stage 1 and Stage 2) and/or Day 8 (Stage 1), until disease progression, maximum benefit, or intolerability.
Arm/Group | Stage 1+Stage 2: GDC-0449 (150 mg) | Stage 1+Stage 2: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg)
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: Average Plasma Concentration at Steady State (Css, Avg) After Multiple Doses of GDC-0449
Description: Steady state GDC-0449 plasma concentrations (Css) were calculated as an average of plasma concentrations from Study Day 21 (Stage 2) or Study Day 28 (Stage 1) onward.
Time Frame: as for outcome 3
Population: PK-evaluable population. Here "number of participants analyzed" = participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mcM
Arm/Group | Stage 1+Stage 2: GDC-0449 (150 mg) | Stage 1+Stage 2: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 38 | 21 | 4 | 15
mcM | 23.1 (10.6) | 19.8 (9.51) | 22.2 (8.38) | 24.5 (6.85)

7. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24) After a Single Dose of GDC-0449
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. Phase I comprised of two stages, a dose-escalation stage with the goal of estimating the maximum tolerated dose (Stage 1), and an expanded cohort to collect additional safety, PK, and PD data at the proposed Phase II dose (Stage 2). Phase II represented the additional cohort initiated with 150 mg hard gelatin capsule identified from the safety, PK and PD data from Stage 1 of the trial.
Time Frame: as for outcome 2
Population: PK-evaluable population.
Measure: Mean (Standard Deviation); unit: mcM*day
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 7 | 9 | 4 | 16
mcM*day
  Phase I | 2.22 (0.966) | 4.24 (1.95) | 4.79 (2.22) | NA (NA) — The arm was only valid for Phase II.
  Phase II | NA (NA) — The arm was only valid for Phase I. | NA (NA) — The arm was only valid for Phase I. | NA (NA) — The arm was only valid for Phase I. | 5.2 (2.79)

8. Primary Outcome: AUC0-24 After Multiple Doses of GDC-0449
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. AUC was estimated if there were extensive PK sampling in more that 50% of the participants to form a curve.
Time Frame: as for outcome 3
Population: AUC0-24 was not reported as there were <50% participants with extensive PK sampling and the PK profiles were flat over 24 hours at steady state which did not allow estimation of AUC0-24.
Arm/Group | Stage 1+Stage 2: GDC-0449 (150 mg) | Stage 1+Stage 2: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg)
Number analyzed (Participants) | 0 | 0 | 0

9. Primary Outcome: Accumulation Index (AI) After Multiple Doses of GDC-0449
Description: AI was calculated using the formula [AI = AUC(0-24) on Day 15/AUC(0-24) on Day 1]. AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. AI was estimated if there were extensive PK sampling in more that 50% of the participants to form a curve.
Time Frame: as for outcome 3
Population: AI was not reported as there were <50% participants with extensive PK sampling and the PK profiles were flat over 24 hours at steady state which did not allow estimation of AI.
Groups:
- Stage 1: GDC-0449: Included participants with any tumor who received a single oral dose of GDC-0449 hard gelatin capsules at a dosage of 150 mg, 270 mg and 540 mg on Day 1. Beginning on Day 8, participants received once daily doses of GDC-0449 150 mg, 270 mg and 540 mg orally, continuing until disease progression, maximum benefit, or intolerability.
Arm/Group | Stage 1: GDC-0449
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants With a Greater Than (>) 2-Fold Down-Modulation of GLI1 Expression in Skin Biopsy-Derived or Hair Follicle-Derived Messenger Ribonucleic Acid (mRNA)
Description: Ribonucleic acid (RNA) was extracted from biopsy specimens of noninvolved skin or hair follicles at baseline and at 7 and 21 days after the start of daily drug therapy. Control mRNA was obtained from formalin-fixed, paraffin-embedded samples of normal skin and hair follicles from participants who were not enrolled in the study.
Time Frame: Baseline up to Day 29
Population: Pharmacodynamic-evaluable population included participants who had hair and/or skin samples available from Day 1 and at least one post-baseline sample while on study treatment. Here "number of participants analyzed" = participants evaluable for this measure and "n"= participants evaluable for the specific category.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: Included all participants from Stage 1 and Stage 2.
Arm/Group | All Participants
Number analyzed (Participants) | 34
percentage of participants
  Skin biopsy (n = 34) | 73.5
  Hair follicle (n = 20) | 30.0

11. Secondary Outcome: Percentage of Participants With a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR): All Participants
Description: BOR was defined as the best objective response (complete or partial response determined by two consecutive investigator assessments which were at least 28 days apart) observed during the treatment period according to RECIST v1.0. CR: disappearance of all target lesions (TLs), with any pathological lymph nodes (whether target or non-target) having a reduction in short axis to less than 10 millimeters (mm). PR: at least a 30 percent (%) decrease in the sum of diameters of TLs, taking as reference the baseline (BL) sum diameters.
Time Frame: Screening, at Week 8 thereafter every 8 weeks, up to Week 116
Population: Efficacy-evaluable population were those with measurable disease at baseline and who received at least 1 dose of GDC-0449 and either had a post-baseline tumor assessment or progressed before any tumor assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma (GDC-0449 [150 mg]) | Stage 2: Basal Cell Carcinoma (GDC-0449 [270 mg]) | Stage 2:Safety Expansion Cohort (GDC-0449 [150 mg]) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 7 | 9 | 4 | 6 | 14 | 10 | 16
percentage of participants | 14.3 | 11.1 | 0.0 | 66.7 | 42.9 | 0.0 | 37.5

12. Secondary Outcome: Percentage of Participants With a BOR of CR or PR: Participants With Basal Cell Carcinoma
Description: BOR was defined as the best objective response observed during the treatment period according to RECIST v1.0. CR: disappearance of all TLs, with any pathological lymph nodes (whether target or non-target) having a reduction in short axis to less than 10 mm. PR: at least a 30% decrease in the sum of diameters of TLs, taking as reference the BL sum diameters.
Time Frame: Screening, at Week 8 thereafter every 8 weeks, up to Week 116
Population: Efficacy-evaluable population; only participants with BCC were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma (GDC-0449 [150 mg]) | Stage 2: Basal Cell Carcinoma (GDC-0449 [270 mg]) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 1 | 1 | 1 | 6 | 14 | 10
percentage of participants | 100.0 | 100.0 | 0.0 | 66.7 | 42.9 | 60.0

13. Secondary Outcome: Duration of Objective Response: All Participants
Description: Duration of response during first line therapy is defined as the time from when response (CR or PR) was first documented to first documented disease progression or death (whichever occurs first) during first line therapy. This was only calculated for participants who achieved a best overall response of CR or PR. Participants who did not progress or die after they had a confirmed response were censored at the date of their last tumor measurement or last follow-up for progression of disease during first line therapy.
Time Frame: Screening, at Week 8 thereafter every 8 weeks, up to Week 116
Population: Efficacy-evaluable population; only participants who achieved a best overall response of CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma (GDC-0449 [150 mg]) | Stage 2: Basal Cell Carcinoma (GDC-0449 [270 mg]) | Stage 2:Safety Expansion Cohort (GDC-0449 [150 mg]) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 1 | 1 | 0 | 4 | 6 | 0 | 6
months | 9.2 [NA to NA] — Upper and lower limits of 95% CI could not be estimated as n=1. | NA [NA to NA] — Median duration of response could not be estimated as median duration of response had not been reached at the time of analysis. |  | 6.1 [3.71 to NA] — Upper limit of CI could not be estimated due to consequence regarding occurrence of events and their censoring. | NA [5.72 to NA] — Median duration of response could not be estimated as median duration of response had not been reached at the time of analysis. |  | 8.3 [3.71 to NA] — Upper limit of CI could not be estimated due to consequence regarding occurrence of events and their censoring.

14. Secondary Outcome: Duration of Objective Response: Participants With BCC
Description: as for outcome 13
Time Frame: Screening, at Week 8 thereafter every 8 weeks, up to Week 116
Population: Efficacy-evaluable participants; only participants with BCC who achieved a best overall response of CR or PR were included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Stage 1+Stage 2: GDC-0449 (150 mg) | Stage 1+Stage 2: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg)
Number analyzed (Participants) | 11 | 7 | 0
months | 8.3 [3.71 to NA] — Upper limit of CI could not be estimated due to consequence regarding occurrence of events and their censoring. | NA [5.72 to NA] — Median duration of response could not be estimated as median duration of response had not been reached at the time of analysis. |

15. Secondary Outcome: Progression-Free Survival (PFS): All Participants
Description: PFS was defined as the time from first dose of GDC-0449 to documented disease progression (deterioration of evaluable lesions and/or tumor-related symptoms defined using RECIST v1.0) or death from any cause within 30 days of the last dose of GDC-0449, whichever occurred first.
Time Frame: Screening, at Week 8 thereafter every 8 weeks, up to Week 116
Population: Efficacy-evaluable population. Number of participants censored for Stage 1 150 mg, 270 mg, and 540 mg were 1, 2, and 1 subjects, respectively and for Stage 2 BCC 150 mg, 270 mg, Stage 2 Safety Expansion Cohort 150 mg, and Stage 2 New Formulation 150 mg were 2, 6, 1, and 6 subjects, respectively.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma (GDC-0449 [150 mg]) | Stage 2: Basal Cell Carcinoma (GDC-0449 [270 mg]) | Stage 2:Safety Expansion Cohort (GDC-0449 [150 mg]) | Stage 2: New Formulation (GDC-0449 [150 mg])
Number analyzed (Participants) | 7 | 9 | 4 | 6 | 14 | 10 | 16
months | 2.0 [0.99 to 14.85] | 1.6 [0.85 to 5.88] | 2.1 [1.25 to 3.02] | 9.6 [5.75 to NA] — Upper limit of CI could not be estimated due to consequence regarding occurrence of events and their censoring. | 12.7 [6.70 to NA] — Upper limit of CI could not be estimated due to consequence regarding occurrence of events and their censoring. | 1.8 [0.76 to 2.10] | 7.1 [0.99 to NA] — Upper limit of CI could not be estimated due to consequence regarding occurrence of events and their censoring.

16. Secondary Outcome: PFS: Participants With BCC
Description: as for outcome 15
Time Frame: Screening, at Week 8 thereafter every 8 weeks, up to Week 116
Population: Efficacy-evaluable population; only participants with BCC were included in the analysis. Number of participants censored for Stage 1+Stage 2 150 mg, and Stage 1+Stage 2 270 mg were 8 and 7 subjects, respectively, and no subject censored from Stage 1 540 mg group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1+Stage 2: GDC-0449 (150 mg) | Stage 1+Stage 2: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg)
Number analyzed (Participants) | 17 | 15 | 1
months | 10.8 [6.67 to NA] — Upper limit of CI could not be estimated due to consequence regarding occurrence of events and their censoring. | 12.7 [6.70 to NA] — Upper limit of CI could not be estimated due to consequence regarding occurrence of events and their censoring. | 1.2 [NA to NA] — Upper and lower limits of 95% CI could not be estimated as n=1.

ADVERSE EVENTS:
Time Frame: From Screening up to 28 days after the last dose of GDC-0449 (Week 116).
Groups:
- Stage 1: GDC-0449 (150 mg): Participants received single dose of GDC-0449 hard gelatin capsules at 150 mg on Day 1, thereafter Day 8 received daily until disease progression, maximum benefit, or intolerability.
- Stage 1: GDC-0449 (270 mg): Stage 1: GDC-0449 (270 mg) Participants received single dose of GDC-0449 hard gelatin capsules at 270 mg on Day 1, thereafter Day 8 received daily dose until disease progression, maximum benefit, or intolerability.
- Stage 1: GDC-0449 (540 mg): Participants received single dose of GDC-0449 hard gelatin capsules at 540 mg on Day 1, thereafter Day 8 received daily dose until disease progression, maximum benefit, or intolerability.
- Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)]: Participants with basal cell carcinoma (BCC) received daily dose of GDC-0449 hard gelatin capsules at 150 mg on Day 1 until disease progression, maximum benefit, or intolerability.
- Stage 2: Basal Cell Carcinoma [GDC-0449 (270 mg)]: Participants with basal cell carcinoma (BCC) received daily dose of GDC-0449 hard gelatin capsules at 270 mg on Day 1 until disease progression, maximum benefit, or intolerability.
- Stage 2:Safety Expansion Cohort [GDC-0449 (150 mg)]: Participants with tolerable safety, pharmacokinetic and pharmacodynamic data from Stage 1 received daily dose of GDC-0449 hard gelatin capsules at 150 mg on Day 1 until disease progression, maximum benefit, or intolerability.
Arm/Group | Stage 1: GDC-0449 (150 mg) | Stage 1: GDC-0449 (270 mg) | Stage 1: GDC-0449 (540 mg) | Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)] | Stage 2: Basal Cell Carcinoma [GDC-0449 (270 mg)] | Stage 2:Safety Expansion Cohort [GDC-0449 (150 mg)] | Stage 2: New Formulation [GDC-0449 (150 mg )]
Serious Adverse Events (participants affected / at risk) | 3/7 | 2/9 | 1/4 | 2/6 | 4/14 | 4/12 | 4/16
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9 | 4/4 | 6/6 | 14/14 | 12/12 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: GDC-0449 (150 mg) (N=7) | Stage 1: GDC-0449 (270 mg) (N=9) | Stage 1: GDC-0449 (540 mg) (N=4) | Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)] (N=6) | Stage 2: Basal Cell Carcinoma [GDC-0449 (270 mg)] (N=14) | Stage 2:Safety Expansion Cohort [GDC-0449 (150 mg)] (N=12) | Stage 2: New Formulation [GDC-0449 (150 mg )] (N=16)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: GDC-0449 (150 mg) (N=7) | Stage 1: GDC-0449 (270 mg) (N=9) | Stage 1: GDC-0449 (540 mg) (N=4) | Stage 2: Basal Cell Carcinoma [GDC-0449 (150 mg)] (N=6) | Stage 2: Basal Cell Carcinoma [GDC-0449 (270 mg)] (N=14) | Stage 2:Safety Expansion Cohort [GDC-0449 (150 mg)] (N=12) | Stage 2: New Formulation [GDC-0449 (150 mg )] (N=16)
Nausea (Gastrointestinal disorders) | 1 | 5 | 1 | 2 | 5 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 4 | 1 | 6
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 2 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 1 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 3 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral cavity fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 4 | 12 | 0 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 1 | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 4 | 0 | 4 | 8 | 6 | 5
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 3 | 2 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 2
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 3
Oedema (General disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1
Chest discomfort (General disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Unevaluable event (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 3 | 1 | 5 | 8 | 2 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Anosmia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Amimia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paresis cranial nerve (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phantom pain (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viith nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 10 | 1 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 1 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 4 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Actinic elastosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Campbell de morgan spots (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 2 | 1 | 4 | 5 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 2 | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Salt craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 5 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 2 | 3 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 3 | 2 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 3 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 3 | 1 | 2 | 4 | 2 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urine (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carbohydrate antigen 19-9 increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram change (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metamyelocyte percentage increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myelocyte percentage increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 1 | 1 | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 4
Depression (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arcus lipoides (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Auricular swelling (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear canal stenosis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.